CLINICAL TRIAL: NCT06623721
Title: Feasibility and Tolerance of Movement-activated Auricular Vagus Nerve Stimulation in Motor Rehabilitation
Brief Title: Movement-activated Auricular Vagus Nerve Stimulation in Rehabilitation
Acronym: sVNS-rehab
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Olivier Lambercy (Other)
Collaborators: Cereneo AG (Industry)
Responsible Party: Sponsor-Investigator, Olivier Lambercy, Adjunct Professor and the Deputy Director of the Rehabilitation Engineering Laboratory at ETH Zurich, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SmartVNSNeuroRehab; 2024-01425 (Registry Identifier: BASEC)
Record Dates: First submitted 2024-09-20; First posted 2024-10-02 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Stroke Rehabilitation; Neurorehabilitation
Keywords: neurorehabilitation; feasibility; vagus; stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Patients undergoing prescribed neurorehabilitation therapy with additional intervention of movement-evoked auricular Vagus nerve stimulation.
  Interventions: Device: Movement-evoked transcutaneous auricular Vagus nerve stimulation

INTERVENTIONS:
Device: Movement-evoked transcutaneous auricular Vagus nerve stimulation — Intervention requires wearing of an inertial measurement unit (IMU) sensor on an affected upper limb together with a transcutaneous auricular Vagus nerve (taVNS) stimulator on an outer ear on the contralateral side.
  Intervention involves IMU measurement-evoked initiation of taVNS during conventional neurorehabilitation therapy that is defined by the patient's doctor and therapist. Typically this is around 60 minutes/day of 50-300 repetitive upper limb movements targeting specific deficits such as flexor synergies and/or wrist, triceps or shoulder activation.
  taVNS intensity is calibrated at the start of every neurorehabilitation session by the patient to the maximal comfortable level with instructions to avoid pain or any serious discomfort. Patient is always accompanied by a therapist trained in the use of taVNS and the device is easy to immediately remove should any discomfort occur.

SUMMARY:
Rehabilitation engineering laboratory (RELab) at the ETH Zurich is recruiting participants with a motor function deficit for studying a novel non-invasive brain stimulation method that may be a promising approach for benefiting motor recovery after conditions like stroke, traumatic brain injury or spinal cord injury. The study will be conducted at the cereneo Hertenstein clinic. Participants with residual motor function deficit due to stroke or spine/brain injury will be undergoing typical neurorehabilitation procedures in addition to the use of the automatically controlled non-invasive Vagus nerve stimulation (taVNS).

This study will analyze the feasibility of this method before it can be used by doctors generally. More specifically, this study aims to test whether controlling taVNS with a wearable wrist-worn sensor during rehabilitation exercises for movement is both practical and safe. This stimulation works by involves sending tiny electric pulses to the outside of the ear after the wrist sensor detects movement. These pulses activate the auricular Vagus nerve and in turn the brain. Over the course of multiple rehabilitation procedures, taVNS may to help with the speed of motor recovery as shown with previous, manually controlled studies. The goal of this study is wants to see if the automatically controlled taVNSs method works well and doesn't cause any harm while people are doing their therapy exercises. If successful, in the future it could offer a new way to improve the recovery process movement for people with motor difficulties.

DETAILED DESCRIPTION:
Transcutaneous auricular vagus nerve stimulation (taVNS) has emerged as a safe and medically approved non-invasive method for stimulating the vagus nerve, utilising a small electrode placed on the outer ear to transcutaneously activate an auricular branch of the vagus nerve. Studies indicate the potential benefits of both invasive and non-invasive vagus nerve stimulation for motor neurorehabilitation, particularly when combined with rehabilitation exercises. A recent pilot study has shown that pairing motor rehabilitation with taVNS in a movement-gated system resulted in improvement on Fugl-Meyer Assessment upper extremity scores and a greater effect size compared to an unpaired taVNS, while administering fewer stimulation pulses. This demonstrates that taVNS paired with movement therapy can reduce the intensity of stimulation, while still producing beneficial results. However, current approaches for performing stimulation during movement require either manual control or complex and non-specific sensor setup. There are no options for tracking and controlling stimulation based on movement kinematics in an objective, unsupervised manner. Therefore, an in-house developed taVNS system will be used (SmartVNS). The system includes inertial measurement unit (IMU) sensors to track patient's movement and then automatically initiates the taVNS stimulation during movements.

The benefit for participants in the study involving transcutaneous auricular vagus nerve stimulation (taVNS) paired with rehabilitation exercises outweighs the potential risks. The intervention, taVNS, is a medically approved procedure with minimal and extremely rare adverse effects, particularly when used within approved parameters. The study protocol ensures that taVNS will be administered at safe and tolerable intensity levels, with immediate removal of electrodes if any discomfort occurs. Additionally, the intervention will not alter the typical rehabilitation program of the participants, and motion-triggered taVNS will be while participants perform repetitive rehabilitation exercise movements with the affected limb. The potential benefits of the study include contributing to the quality of future neurorehabilitation outcomes and informing decisions for protocols in future clinical studies to explore the efficacy of taVNS in enhancing neurorehabilitation and motor learning in adults with motor deficits. Overall, the study aims to prioritise participant safety while offering the potential for meaningful therapeutic benefits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ability to follow study instructions
* At least 1-2 weeks after a stroke or traumatic brain/spinal cord injury and with a residual motor deficit.

Exclusion Criteria:

* Inability to give informed consent or understand the tasks, other neurological or psychiatric illness that could confound execution/recovery. E.g. Global inattention or receptive aphasia.
* Presence of ongoing dysphagia or aspiration difficulties
* Subject receiving medication that may significantly interfere with actions of taVNS on neurotransmitter systems at study enrollment
* Prior injury to vagus nerve, either bilateral or unilateral (e.g., injury during carotid endarterectomy)
* Severe depression (Beck Depression Scale > 29)
* Current use of any implanted electronic device, such as a pacemaker or other neurostimulator
* Medical or mental instability (diagnosis of personality disorder, psychosis, or substance abuse) that would prevent the subject from meeting protocol timeline
* Pregnancy or plans to become pregnant or to breastfeed during the study period
* Current requirement, or likely future requirement, of diathermy during the study duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-10-03 (Estimated); Study Completion 2025-10-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of automatic movement-initiated taVNS | From enrollment to the end of treatment at 2 or at 4 weeks with an additional follow-up at 1 week after
  Perceived feasibility of automatic movement-initiated taVNS, assessed through validated questionnaires. This includes subjective ratings on ease of use, comfort, and perceived effects by therapists and patients. Questionnaires include: UMUX, IMI and UE.

SECONDARY OUTCOMES:
Feasibility of automatic movement detection during therapy | On the first and last sessions of the study at weeks 1 and 2 or 4.
  Agreement between manual movement detection by therapists and automatic sensor-triggered stimulation timings, based on ground-truth video recording, assessing technical feasibility.
Tolerance and safety | From enrollment to the end of treatment at 2 or at 4 weeks.
  Recording incidences of adverse events and subjective unstructured feedback.
Motor deficit | From enrollment to the end of treatment at 2 or at 4 weeks.
  Analysis of routine clinical assessments of motor deficit using the Fugl-Meyer Assessment for upper extremity (FMA-UE). Higher FMA-UE scores indicate reduction of deficit and improvement in patient's motor skills. Comparison of post-rehabilitation against baseline to ensure no deterioration, using statistical comparison of evaluation of standard clinical assessments performed during patients stay.
Mood assessment | From enrollment to the end of treatment at 2 or at 4 weeks.
  Description: Analysis of routine clinical assessments of assessning mood by using the Hospital Anxiety and Depression Scale (HADS). High scores indicate abnormal anxiety and/or depression. Comparison of post-rehabilitation against baseline to ensure no deterioration, using statistical comparison of evaluation of standard clinical assessments performed during patients stay.
  Time Frame: From enrollment to the end of treatment at 2 or at 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Cereneo Hertenstein, Weggis, Switzerland

IPD SHARING:
Plan to Share IPD: No
Not planned.

REFERENCES:
- [Background] Badran BW, Peng X, Baker-Vogel B, Hutchison S, Finetto P, Rishe K, Fortune A, Kitchens E, O'Leary GH, Short A, Finetto C, Woodbury ML, Kautz S. Motor Activated Auricular Vagus Nerve Stimulation as a Potential Neuromodulation Approach for Post-Stroke Motor Rehabilitation: A Pilot Study. Neurorehabil Neural Repair. 2023 Jun;37(6):374-383. doi: 10.1177/15459683231173357. Epub 2023 May 20. PMID 37209010
- [Background] Baig SS, Kamarova M, Bell SM, Ali AN, Su L, Dimairo M, Dawson J, Redgrave JN, Majid A. tVNS in Stroke: A Narrative Review on the Current State and the Future. Stroke. 2023 Oct;54(10):2676-2687. doi: 10.1161/STROKEAHA.123.043414. Epub 2023 Aug 30. PMID 37646161
- [Background] Dawson J, Liu CY, Francisco GE, Cramer SC, Wolf SL, Dixit A, Alexander J, Ali R, Brown BL, Feng W, DeMark L, Hochberg LR, Kautz SA, Majid A, O'Dell MW, Pierce D, Prudente CN, Redgrave J, Turner DL, Engineer ND, Kimberley TJ. Vagus nerve stimulation paired with rehabilitation for upper limb motor function after ischaemic stroke (VNS-REHAB): a randomised, blinded, pivotal, device trial. Lancet. 2021 Apr 24;397(10284):1545-1553. doi: 10.1016/S0140-6736(21)00475-X. PMID 33894832